CLINICAL TRIAL: NCT00355472
Title: Phase I Dose Escalation Study of KW-0761 in Patients With Relapsed Adult T-Cell Lymphoma (ATL) and Peripheral T-Cell Lymphoma (PTCL)
Brief Title: Phase I Study of KW-0761 in Relapsed Patients With CCR4-Positive ATL and PTCL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0761-0501
Record Dates: First submitted 2006-07-20; First posted 2006-07-24 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Adult T-Cell Leukemia and Lymphoma (ATL); Adult Peripheral T-Cell Lymphoma (PTCL)
Keywords: Adult T-Cell Leukemia; ATL; Adult Peripheral T-Cell Lymphoma; PTCL
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell; Lymphoma, T-Cell, Peripheral | interventions — mogamulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): KW-0761
  Interventions: Drug: KW-0761

INTERVENTIONS:
Drug: KW-0761 — IV administration at 4 escalating dose levels.

SUMMARY:
This is a Phase I label dose escalation study of KW-0761 in relapsed patients with CCR4 positive Adult T-Cell Leukemia-Lymphoma (ATL) and Peripheral T-Cell lymphoma (PTCL).

DETAILED DESCRIPTION:
This is a Phase I open-label dose escalation study of KW-0761 in relapsed patients with CCR4 positive Adult T-Cell Leukemia-Lymphoma (ATL) and Peripheral T-Cell Lymphoma (PTCL). This study is designed to evaluate safety, pharmacokinetics, immunogenicity and preliminary efficacy. Enrollment will proceed until a maximum tolerated dose (MTD) and a recommended Phase II dose (RPIID) have been established.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of a CCR4-positive ATL and PTCL that is any of the following:

A. ATL (Adult T-Cell Leukemia-Lymphoma)

* Seropositive for anti-Human T-lymphotrophic Virus type-I (HTLV-I) antibody;
* Acute, Lymphoma, or Chronic phase with high-risk factors (within 14 days before the study entry);

B. PTCL (Peripheral T-Cell Lymphoma)

* Includes Mycosis Fungoides and Sezary Syndrome;

  2: Relapsed to the latest standard chemotherapy;

  3: Received at least one prior chemotherapy;

  4: After 4 weeks from a prior therapy;

  5: Have measurable disease;

  6:Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1;

  7: Male or female, at least 20 years and not older than 70 years of age;

  8: Signed written informed consent;

  9: Stay in hospital for 4 weeks;

  10: HBs antigen: negative, HBV-DNA: below the limit of quantification (within 14 days before the study entry);

  11: Adequate bone marrow, hepatic and cardiac function including the followings:
* Neutrophil count ≥ 1,500 /mm3,
* Platelets ≥ 75,000 /mm3,
* Hemoglobin ≥ 8.0 g/dL
* Serum creatinine ≤ 1.5 x ULN;
* Serum SGOT (AST) and SGPT (ALT) ≤ 2.5 x ULN (≤ 5.0 x ULN if considered due to disease involvement in liver);
* Serum bilirubin ≤ 1.5 x ULN (≤ 3.0 x ULN if considered due to disease involvement in liver)
* Serum calcium ≤ 11.0 mg/dL
* PaO2 ≥ 65 mmHg or SaO2 ≥ 90%
* No clinically significant Electrocardiogram abnormality
* Left Ventricular Ejection Fraction ≥ 50% [by ECHO or MUGA]

Exclusion Criteria:

1. Co-existing active infection or any co-existing medical condition that may compromise the safety of patients during the study, affect the patient's ability to complete the study, or interfere with interpretation of study results;
2. Active tuberculosis;
3. Prior stem cell transplantation;
4. Myocardial infarction (within 12 months prior to the study entry);
5. Concurrent acute or chronic hepatitis, or cirrhosis;
6. Anti-HCV: positive, Anti-HIV: positive
7. Concurrent active malignant disease;
8. Known allergic reaction to antibody therapy;
9. Concomitant treatment with systemic steroids;
10. Prior and Concurrent psychiatric disorder including dementia, epilepsy or any other CNS diseases;
11. Evidence of CNS metastasis at baseline;
12. Prior and Concurrent spinal cord disease;
13. Radiation therapy for bulky mass disease at the time of study entry or considered to require radiation therapy during the study;
14. Female patients who are pregnant or breast feeding;
15. Female patients of childbearing potential, unwilling to use an approved, effective means of contraception in accordance with the institution's standards;
16. Treatment with any other investigational agent within the 4 months prior to study entry;
17. For any reason is judged by the Investigator to be inappropriate for study participation, including an inability to communicate or cooperate with the Investigator.

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Kyowa Kirin Co., Ltd.
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Background] Ishida T, Ueda R. CCR4 as a novel molecular target for immunotherapy of cancer. Cancer Sci. 2006 Nov;97(11):1139-46. doi: 10.1111/j.1349-7006.2006.00307.x. Epub 2006 Sep 5. PMID 16952304
- [Background] Yano H, Ishida T, Inagaki A, Ishii T, Ding J, Kusumoto S, Komatsu H, Iida S, Inagaki H, Ueda R. Defucosylated anti CC chemokine receptor 4 monoclonal antibody combined with immunomodulatory cytokines: a novel immunotherapy for aggressive/refractory Mycosis fungoides and Sezary syndrome. Clin Cancer Res. 2007 Nov 1;13(21):6494-500. doi: 10.1158/1078-0432.CCR-07-1324. PMID 17975162
- [Background] Yano H, Ishida T, Inagaki A, Ishii T, Kusumoto S, Komatsu H, Iida S, Utsunomiya A, Ueda R. Regulatory T-cell function of adult T-cell leukemia/lymphoma cells. Int J Cancer. 2007 May 1;120(9):2052-7. doi: 10.1002/ijc.22536. PMID 17278106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 6 February 2007 through 22 October 2008
Groups:
- KW-0761: KW-0761 was administered 4 times at one-week intervals at a dose of 0.01, 0.1, 0.5 or 1.0 mg/kg in patients with CC chemokine 4 receptor (CCR4) positive Adult T-Cell Leukemia-Lymphoma (ATL) or CCR4 positive Peripheral T-Cell Lymphoma (PTCL)
Period: Overall Study
Arm/Group | KW-0761
Started | 16
Completed | 15
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- KW-0761: KW-0761 was administered 4 times at one-week intervals at a dose of 0.01, 0.1, 0.5 or 1.0 mg/kg in patients with CCR4 positive ATL or CCR4 positive PTCL
Arm/Group | KW-0761
Number analyzed (Participants) | 16
Age Continuous [Median (Full Range); unit: years] | 62 [46 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Diagnosis [Number; unit: participants]
  ATL | 13
  PTCL | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-Limiting Toxicities (DLTs)
Description: Subjects who were properly monitored for DLTs were to be analyzed to determine the number of subjects with a DLT by dose level.
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | KW-0761
Number analyzed (Participants) | 16
participants | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The dose level at which Dose-Limiting Toxicity (DLT) was recognized was to be regarded as Maximum Tolerated Dose (MTD), and the dose level below MTD by one level was to be regarded as the recommended dose level (when MTD was not reached, 1.0 mg/kg was to be regarded as the recommended dose level) and 3 more subjects were to be newly added to the recommended dose level.
Time Frame: 28 days
Measure: Number; unit: mg/kg
Arm/Group | KW-0761
Number analyzed (Participants) | 16
mg/kg | 1.0

3. Secondary Outcome: Antitumor Effect
Description: The antitumor response criteria (Complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD)) were created based on the criteria for non-Hodgkin's lymphoma and chronic lymphocytic leukemia provided in the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology as well as the criteria for non-Hodgkin's lymphoma by the Lymphoma Study Group of the Japan Clinical Oncology Group (JCOG-LSG).
Time Frame: 50 days
Measure: Number; unit: participants
Groups:
- KW-0761 0.01mg; KW-0761 0.1mg; KW-0761 0.5mg; KW-0761 1.0mg: IV infusions of KW-0761 once/week for 4 weeks
Arm/Group | KW-0761 0.01mg | KW-0761 0.1mg | KW-0761 0.5mg | KW-0761 1.0mg
Number analyzed (Participants) | 3 | 4 | 3 | 6
participants
  Complete Response (CR) | 0 | 1 | 0 | 1
  Uncertain Complete Response (CRu) | 0 | 0 | 0 | 0
  Partial Response (PR) | 1 | 0 | 0 | 2
  Stable Disease (SD) | 1 | 2 | 0 | 2
  Progressive Disease (PD) | 1 | 1 | 3 | 1
  Not Evaluable (NE) | 0 | 0 | 0 | 0

4. Primary Outcome: Pharmacokinetics-Plasma KW-0761 Concentrations
Description: Plasma KW-0761 concentrations were to be summarized in tabular form with the descriptive statistics on a dose-by-dose basis. Individual and mean (+ standard deviation) plasma KW-0761 concentrations on an actual or logarithmic scale were to be plotted against the time of blood sampling.
Time Frame: 0-7 days post final dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | KW-0761 0.01mg | KW-0761 0.1mg | KW-0761 0.5mg | KW-0761 1.0mg
Number analyzed (Participants) | 3 | 4 | 3 | 6
ng/mL
  Cmax | 350.0 (47.8) | 2806.7 (1664.5) | 15181.2 (872.0) | 40428.4 (5350.8)
  Ctrough | 158.2 (7.4) | 1515.2 (1873.4) | 6824.7 (872.9) | 19516.8 (4264.7)

5. Primary Outcome: Pharmacokinetics-Pharmacokinetic Parameters of KW-0761 (AUC0-7 Days)
Description: The pharmacokinetic parameters of the subjects were to be individually calculated, and their descriptive statistics were to be calculated on a dose-by-dose basis.
Time Frame: 0-7 days post final dose
Population: AUC0-7 days
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | KW-0761 0.01mg | KW-0761 0.1mg | KW-0761 0.5mg | KW-0761 1.0mg
Number analyzed (Participants) | 3 | 4 | 3 | 6
ng·h/mL | 36586 (2987) | 327609 (322298) | 1625609 (142277) | 4190238 (544757)

6. Primary Outcome: Pharmacokinetics-Pharmacokinetic Parameters of KW-0761 (t1/2)
Description: as for outcome 5
Time Frame: 0 to 28 days post final dose and follow-up examinations (1 month and 2 months after the end of the post-dosing observation period).
Population: t1/2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | KW-0761 0.01mg | KW-0761 0.1mg | KW-0761 0.5mg | KW-0761 1.0mg
Number analyzed (Participants) | 3 | 4 | 3 | 6
hours | 179 (40) | 201 (196) | 332 (122) | 462 (51)

7. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the period from the day starting the first KW-0761 dosing to the day of PD identification (or the day of death if the subject died before PD was documented). Subjects were to be censored at the time of starting post-treatment, if it was started before PD identification.
Time Frame: Baseline to response
Measure: Median (Full Range); unit: days
Arm/Group | KW-0761
Number analyzed (Participants) | 16
days | 46.5 [8 to 617]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | KW-0761 0.01mg | KW-0761 0.1mg | KW-0761 0.5mg | KW-0761 1.0mg
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KW-0761 0.01mg (N=3) | KW-0761 0.1mg (N=4) | KW-0761 0.5mg (N=3) | KW-0761 1.0mg (N=6)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KW-0761 0.01mg (N=3) | KW-0761 0.1mg (N=4) | KW-0761 0.5mg (N=3) | KW-0761 1.0mg (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Infusion-related reaction (General disorders) | 3 (3) | 3 (3) | 3 (3) | 4 (4)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 4 (4) | 3 (3) | 6 (6)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2) | 3 (3) | 4 (4)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 2 (2) | 3 (3) | 4 (4)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophil percentage increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Platelet function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other